CLINICAL TRIAL: NCT05752318
Title: APRIL Study: Analysis of the Persistence, Reservoir and HIV Latency
Brief Title: Analysis of the Persistence, Reservoir and HIV Latency
Acronym: APRIL
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8825
Record Dates: First submitted 2023-01-12; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-01

CONDITIONS: HIV Infected Individuals; Informed Consent
Keywords: HIV; Reservoir; Latency; Persistence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The APRIL study aims at analyzing HIV reservoirs, latency and persistence on antiretroviral therapy. It enrolls HIV-infected adults providing blood samples of which peripheral blood mononuclear cells are stored. The frequency, phenotype and inducibility of HIV-infected cells are then analyzed. These parameters may vary across the different clinical and therapeutic settings.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infection
* Adults (>18 years)
* Social insurance
* Informed consent

Exclusion Criteria:

* HIV-uninfected
* <18 years
* Lack of social insurance
* Lack or withdraw of consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: HIV-infected adults
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-02-27 (Estimated); Primary Completion 2027-01-25 (Estimated); Study Completion 2027-02-25 (Estimated)

PRIMARY OUTCOMES:
HIV-Flow | 1 day